CLINICAL TRIAL: NCT06461247
Title: Compliance With Standard Care vs Ready to Eat Meals Prior to Bariatric Surgery - a Randomised Controlled Trial
Brief Title: Compliance With Standard Care vs Ready to Eat Meals Prior to Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/00240
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Bariatric Surgery Candidate
Keywords: Weight loss; Very Low Calorie Diet; Body Weight
MeSH Terms: conditions — Weight Loss; Body Weight | interventions — Meals

STUDY DESIGN:
Intervention Model Description: Standard Care Group (n=70): Participants will be having liquid meal replacement for breakfast, lunch, and dinner for 4 weeks. Additionally, patients are to prepare 1 serving of non-starchy vegetables are to be included for lunch and dinner.
  Intervention Group (n=70): Participants will be provided with VLCD RTE meals for lunch and dinner for 4 weeks and advised on a healthy keto breakfast.
  Both groups will be recommended to keep within the calorie limit to 800kcal and 50g net carbohydrates per day.
Masking Description: It is not feasible to apply blinding to the study design due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very Low Calorie Diet Ready-to-eat (VLCD RTE) meals (Experimental): Participants (n=70) in the VLCD RTE meals group will be advised to follow a calorie-restricted healthy ketogenic diet , consuming a maximum of 800 calories and 50g net carbohydrate intake daily.
  Participants will be provided with VLCD RTE meals for lunch and dinner for 4 weeks and advised on a healthy keto breakfast.
  The participants will be expected to self-monitor their weight, physical activity and diet logs via the nutritionist buddy keto app. There will be in app virtual reminders (automated and by dietitians via the chat function) sent via the nutritionist buddy keto application for the 1 month for participants to log in their weight and meals.
  Interventions: Other: Very Low Calorie Diet Ready-to-eat (VLCD RTE) meals
- Liquid Meal Replacement (Active Comparator): Participants (n=70) in the liquid meal replacement group will be advised to follow very low-calorie diet, with a maximum of 800 calories and 50g net carbohydrate intake daily.
  Participants will be provided with a liquid meal replacement for breakfast, lunch, and dinner for 4 weeks. Additionally, patients are to prepare 1 serving of non-starchy vegetables are to be included for lunch and dinner.
  The participants will be expected to self-monitor their weight, physical activity and diet logs via the nutritionist buddy keto app. There will be in app virtual reminders (automated and by dietitians via the chat function) sent via the nutritionist buddy keto application for the 1 month for participants to log in their weight and meals.
  Interventions: Other: Standard Care Group

INTERVENTIONS:
Other: Very Low Calorie Diet Ready-to-eat (VLCD RTE) meals — Participants will be provided with VLCD RTE meals for lunch and dinner for 4 weeks and advised on a healthy ketogenic breakfast. Participant will be expected to adhere to VLCD regimen containing 800 calories per day or fewer and keep within 50g net carbohydrates a day.
  Arms: Very Low Calorie Diet Ready-to-eat (VLCD RTE) meals
Other: Standard Care Group — Participants will be provided with liquid meal replacement for breakfast, lunch, and dinner for 4 weeks. Additionally, patients are to prepare 1 serving of non-starchy vegetables are to be included for lunch and dinner. Participant will be expected to adhere to VLCD regimen containing 800 calories per day or fewer and keep within 50g net carbohydrates a day.
  Arms: Liquid Meal Replacement

SUMMARY:
Currently, a ketosis-inducing programme, usually a liquid meal replacement, is the standard of care for pre-operative dietary management. However, compliance with liduiqd meal replacement is challenging primarily due to individual taste preferences, limited variety, having to take a liquid diet, lifestyle factors, and other obstacles. Therefore, there is a need for RTE meals to enhance patient satisfaction and compliance, ultimately resulting in improved pre-operative weight loss outcomes. Hence, this RCT study aims to determine whether Very Low Calorie Diet Ready-to-eat (VLCD RTE) meals would lead to greater compliance as measured by blood ketones and meal logging via Nutritionist Buddy app (nBuddy App) compared to standard care liquid meal replacement (Optifast) prior to bariatric surgery.

DETAILED DESCRIPTION:
The obesity rate in Singapore is rising, mirroring a similar worrying global trend. Bariatric surgery has been the only long-term method proven to overcome severe obesity and it has become an increasingly common and effective treatment option. Preoperative weight loss is required to reduce cardiovascular risk, liver volume and decrease intra-abdominal fat. This leads to enhanced surgical visibility and surgical access resulting in reduced intra- and postoperative complications.

Currently, a ketosis-inducing programme, usually a liquid meal replacement, is the standard of care for pre-operative dietary management. However, compliance with liquid meal replacement is challenging primarily due to individual taste preferences, limited variety, having to take a liquid diet, lifestyle factors, and other obstacles. It was found for taste and gastrointestinal side effects to be the main issues.

Therefore, RTE meals are carefully formulated to provide the calculated calorie, controlled net carbohydrate content, and are low in saturated and trans fat. By incorporating these meals as a VLCD diet regime, it would allow patients to still enjoy the chewing sensation and local favourites and flavours, while enjoying mealtime with their friends and families.

In this randomised controlled trial, patients listed for bariatric surgery from the NUH Weight Management Clinic in Singapore will undergo randomization into either the Standard Care or Intervention group during the baseline visit.

* Standard Care Group (n=70): Participants will be provided with liquid meal replacements for breakfast, lunch, and dinner for 4 weeks. Additionally, patients are to prepare 1 serving of non-starchy vegetables are to be included for lunch and dinner.
* Intervention Group (n=70): Participants will be provided with the VLCD RTE meals for lunch and dinner for 4 weeks and advised on a healthy keto breakfast.

All eligible participants (n=140) will be advised to keep within the 800 calorie limit and 50g net carbohydrate limit per day. They will receive guidance from a dietitian on lifestyle changes and pre-bariatric surgery VLCD diets. Participants in both groups will also be advised to download the nutritionist Buddy Keto app for monitoring of compliance, food intake, steps count, weight progress and in app virtual reminders (automated and by dietitians via the chat function).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 to 65 years old
* Scheduled for bariatric surgery at least 1 month prior
* BMI ≥ 27.5 kg/m2 (with type 2 diabetes mellitus or metabolic syndrome)
* Owns a smart phone with data plan
* English speaking

Exclusion Criteria:

* Cognitive impairment.
* Hypothyroidism
* Chronic kidney disease
* Hypothyroidism
* Depression with ongoing psychology follow up
* Type 1 diabetes
* Liver Cirrhosis
* Pregnancy
* Heart Failure
* Active cancer or in remission for less than 5 years
* Vegetarian
* Observing the fast during the month of Ramadan
* Undergoing treatment with anti obesity medications (eg: Phentermine/Orlistat/Contrave/GLP-1 analogues etc)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Compliance rate of the RTE meals | Daily for intervention period of 28 days
  The compliance rate is assessed via food logging in the nutritionist buddy keto app
Blood Ketones Measurement | 1st week, 2nd week, 3rd week, 4th week, surgery day
  Fasting blood ketone measurements measured at study visit

SECONDARY OUTCOMES:
Satisfaction of the RTE meals | 3rd week and surgery day
  Assessed via a self-reported questionnaire with a numeric scale of 1 to 5
Weight Change | 1st week, 2nd week, 3rd week, 4th week, surgery day
  Weight changes at study visit

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Tay, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - Alexandra Hospital, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will remain confidential and only accessible via lock and keys by the researchers.